CLINICAL TRIAL: NCT04525365
Title: Pleural Suction and Evacuation in the Moment of Thoracostomy Tube Procedure in Traumatic Hemothorax Patients: A Randomized Study
Brief Title: Pleural Suction Additional to Thoracostomy Tube for Traumatic Hemothorax
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not possible to achieve adequate recruitment to complete the necessary sample. The rate at which patients are recruited does not allow for continued participation
Sponsor: Hospital Pablo Tobón Uribe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017.019
Record Dates: First submitted 2020-06-11; First posted 2020-08-25 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Traumatic Hemothorax
MeSH Terms: interventions — Thoracentesis

STUDY DESIGN:
Intervention Model Description: Pleural suction under sedation vs Tube Thoracostomy without pleural suction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pleural aspiration (Experimental): Pleural aspiration under sedation
  Interventions: Procedure: Pleural aspiration
- Closed Thoracostomy (Active Comparator): Actual management
  Interventions: Procedure: Pleural aspiration

INTERVENTIONS:
Procedure: Pleural aspiration — Pleural aspiration
  Other Names: Closed Thoracostomy

SUMMARY:
The primary treatment for traumatic hemothorax, is a thoracostomy tube. Some of these patients develop a clotted hemothorax by insufficient drainage. This complication needs surgical resolution and can generate an empyema. One strategy to reduce this complication is pleural suction under sedation before the thoracostomy tube. The aim of the study is define if the procedure really lower the incidence of clotted hemothorax. The investigators design and open label, randomized, interventional study, comparing the realization of the pleural suction and thoracostomy tube alone

DETAILED DESCRIPTION:
Traumatic hemothorax is a common emergency and is commonly the result of trauma, both blunt and penetrating. Although closed drainage thoracostomy is commonly adequate for the initial management of a hemothorax in most cases, failure of the closed thoracostomy and formation of clotted hemothorax can occur in up to 5 to 30% of cases. This complication requires surgical treatment and can generate an empyema, which is a serious infection.

Therefore, the investigators want to impact through a simple and low-cost procedure such as traumatic hemothorax aspiration in the adult population, prior to insertion and fixation of the thoracostomy tube under sedation, to evacuate all the hemothorax present, thus reducing the formation of clots in these patients, and the probability of clotted hemothorax.

Methods: Initially, all patients with penetrating or closed chest trauma that came to the emergency department, are evaluated clinically and with a chest x-ray. With this information, the investigators diagnose patients with traumatic hemothorax or hemopneumothorax, and if is a candidate for drainage with closed thoracostomy. The patient will receive a dose of prophylactic antibiotic, which will be 2 gr of first-generation Cephalosporin, or 600mg iv of Clindamycin for patients allergic to penicillin. At the time of performing the closed thoracostomy procedure, and after approval and signing of the informed consent for the study by the patient or his family member in charge, a consecutive number is assigned with prior randomization of each of the groups in EPIDAT 4.0. In case of being an intervention group, a superficial sedation of the patient will be carried out in the emergency department. Moderate sedation or conscious sedation is performed. The pleura is opened and a sterile adult Yankauer plastic suction cannula (Plus-vital, CE0197, Greetmed RPC) is inserted with closed suction. The cannula will be directed towards the posterior costodiaphragmatic recess at which point hemothorax aspiration will begin at -80 cubic centimeters of water (ccH2O) until complete evacuation is achieved. At the end of the suction, the hemithorax cannula is removed and a silicone 32 French (Fr) thoracostomy tube is inserted, which is subsequently fixed with a non-absorbable 0-gauge suture. The chest tube is connected to a 3-bottle thoracic drainage system ( Oasis Dry suction Water seal 3600 single collection) without continuous pleural suction. After the procedure, a control chest X-ray will be performed within 3 hours to verify the position of the tube, hemothorax drainage, and lung expansion. The clinical and radiological follow up, will be made by surgeon criteria, until the patient develop a clotted hemothorax or is discharged. The investigators will follow this patients by phone after a month. Description and treatment of any adverse events will be made.

Analysis of each of the variables will be carried out in the two groups. Chi2 test to establish statistical significance of these differences, with a bivariate analysis.

Registry of data will be made by the investigators, the source will be the clinical records, and the month phone call, will be made by secondary investigators.

Sample size is of 250 participants, and is planned for 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic hemothorax that needs a Thoracostomy tube procedure

Exclusion Criteria:

* Previous hemothorax in the same hemithorax
* Hemodynamic instability
* Massive hemothorax
* Obtaining saliva, bile, intestinal or gastric material, chyle at the time of performing the procedure
* Closed thoracostomy performed in other institution
* Need of mayor surgical intervention in thorax
* Contraindication for sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2024-03-05 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Clotted hemothorax | One month
  Rate of clotted hemothorax found after Thoracostomy tube procedure or pleural aspiration procedure
Empyema | One month
  Rate of empyema found after Thoracostomy tube procedure

SECONDARY OUTCOMES:
Pleural aspiration procedure complications | One month
  Describe the percentage of patients with complications associated with the pleural aspiration procedure in patients scheduled for thoracostomy tube procedure

CONTACTS AND LOCATIONS:
Overall Officials: Willfredy Castano, MD, Principal Investigator — Pablo Tobon Uribe Hospital, Thoracic Surgeon
Locations (1):
- Pablo Tobon Uribe Hospital, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No
We not consider to share the participant data by laws in our country

REFERENCES:
- [Background] Ramanathan R, Wolfe LG, Duane TM. Initial suction evacuation of traumatic hemothoraces: a novel approach to decreasing chest tube duration and complications. Am Surg. 2012 Aug;78(8):883-7. PMID 22856496
- [Background] Karmy-Jones R, Holevar M, Sullivan RJ, Fleisig A, Jurkovich GJ. Residual hemothorax after chest tube placement correlates with increased risk of empyema following traumatic injury. Can Respir J. 2008 Jul-Aug;15(5):255-8. doi: 10.1155/2008/918951. PMID 18716687
- [Background] Bradley M, Okoye O, DuBose J, Inaba K, Demetriades D, Scalea T, O'Connor J, Menaker J, Morales C, Shiflett T, Brown C. Risk factors for post-traumatic pneumonia in patients with retained haemothorax: results of a prospective, observational AAST study. Injury. 2013 Sep;44(9):1159-64. doi: 10.1016/j.injury.2013.01.032. Epub 2013 Feb 19. PMID 23433600
- [Background] DuBose J, Inaba K, Demetriades D, Scalea TM, O'Connor J, Menaker J, Morales C, Konstantinidis A, Shiflett A, Copwood B; AAST Retained Hemothorax Study Group. Management of post-traumatic retained hemothorax: a prospective, observational, multicenter AAST study. J Trauma Acute Care Surg. 2012 Jan;72(1):11-22; discussion 22-4; quiz 316. doi: 10.1097/TA.0b013e318242e368. PMID 22310111
- [Background] Villegas MI, Hennessey RA, Morales CH, Londono E. Risk factors associated with the development of post-traumatic retained hemothorax. Eur J Trauma Emerg Surg. 2011 Dec;37(6):583-9. doi: 10.1007/s00068-010-0064-3. Epub 2010 Dec 4. PMID 26815469

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT04525365/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT04525365/ICF_001.pdf